CLINICAL TRIAL: NCT04001179
Title: Exploratory Metabolomics Study of Exhaled Breath in Pulmonary Embolism
Acronym: MetabolAir
Status: Terminated | Type: Observational
Why Stopped: recruitment difficulties
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7252
Record Dates: First submitted 2019-06-20; First posted 2019-06-27 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2023-08

CONDITIONS: Pulmonary Embolism
Keywords: Early diagnosis; Mass spectrometry; Volatile Organic Compounds; Metabolomics; Breath Tests; Biomarkers
MeSH Terms: conditions — Pulmonary Embolism; Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Exhaled breath (volatile organic compounds trapped on polymer cartridges)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Presence of pulmonary embolism: ≥ 1 noninfused and normoventilated segment(s) by pulmonary tomoscintigraphy
  Interventions: Other: Pulmonary embolism diagnosis by nuclear medicine imaging
- No pulmonary embolism: Pulmonary perfusion without anomaly (segmental or sub-segmental) by pulmonary tomoscintigraphy
  Interventions: Other: Pulmonary embolism diagnosis by nuclear medicine imaging

INTERVENTIONS:
Other: Pulmonary embolism diagnosis by nuclear medicine imaging — nuclear medicine imaging

SUMMARY:
Pulmonary embolism is a frequent and recurrent pathology, especially in the elderly. It is often preventable, with high mortality and morbidity, making it a major public health issue. The clinical presentation of pulmonary embolism is non-specific and very highly variable, ranging from asymptomatic thrombus diagnosed incidentally to sudden death. The current diagnosis of pulmonary embolism is based on several diagnostic techniques, mainly non-invasive, which should be used sequentially.

We propose to sample the volatile organic compounds using a device that allows them to be trapped on polymer cartridges. Sampling will be performed under monitoring of respiratory pressure and a capnograph to collect alveolar and upper respiratory tract air separately without contamination of the oral cavity or sinuses.

This exploratory metabolic analysis will be non-targeted (analysis of all molecules detectable without a priori).

The main objective of the study is to identify specific metabolic profiles to predict the results of ventilation-perfusion pulmonary tomoscintigraphy in subjects undergoing this examination for suspected acute pulmonary embolism.

Secondary purposes :

* To identify metabolic profiles to be used to predict, in combination with clinical probability scores, the results of ventilation-perfusion pulmonary tomoscintigraphy in subjects undergoing this examination for suspected acute pulmonary embolism.;
* To correlate metabolic profiles with the topography of embolized lung territories

ELIGIBILITY:
Inclusion Criteria:

* Male or female, at least 18 years old
* Patients with clinical suspected pulmonary embolism
* Patient willing and able to provide informed consent

Exclusion Criteria:

* Contraindications to pulmonary ventilator-perfusion tomoscintigraphy
* All types of thrombolytic or anticoagulant treatment
* Diagnosis of pulmonary embolism established prior to inclusion in the study
* Massive pulmonary embolism (systolic pressure < 90 mm Hg)
* Pregnancy
* Breastfeeding

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients presenting to the Nuclear Medicine Department of our hospital for a pulmonary ventilation-perfusion tomoscintigraphy will be proposed to participate in the study
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
quantitative comparison of metabolic profiles | Metabolites are collected immediately before pulmonary tomoscintigraphy
  The quantitative variables compared between the two "contributive" groups are the relative quantities of volatile organic compounds (metabolites) detected by chromatographic techniques coupled with mass spectrometry in exhaled air samples.

SECONDARY OUTCOMES:
Wells score or revised Geneva score | Clinical scores are collected immediately before pulmonary tomoscintigraphy
  The first secondary outcome consists of the primary outcome (quantitative metabolic variables) to which are added quantitative variables of clinical probability score for pulmonary embolism (Wells score or revised Geneva score).
number and location of deficient segments on ventilation-perfusion pulmonary tomoscintigraphy. | day 1
  number and location of deficient segments on ventilation-perfusion pulmonary tomoscintigraphy.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Agin, PhD, Principal Investigator — University Hospital, Strasbourg, France
Locations (1):
- University Hospital, Strasbourg, france, Strasbourg, France